CLINICAL TRIAL: NCT04956146
Title: A Single Arm,Open-label, Study of Fruquintinib Combined With Sintilimab and Chemotherapy in Patients With Unresectable or Metastatic Advanced Wild-type Genotype Non-squamous Non-small Cell Lung Cancer
Brief Title: Fruquintinib Combined With Sintilimab and Chemotherapy in the Treatment of Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-L101
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib Combined With Sintilimab and Chemotherapy (Experimental)
  Interventions: Drug: Fruquintinib，Sintilimab，Pemetrexed，Carboplatin

INTERVENTIONS:
Drug: Fruquintinib，Sintilimab，Pemetrexed，Carboplatin — Fruquintinib,fruquintinib at the dose determined in phase safety lead-in,5mg-intermittent (2 weeks on/ 1 week off) ，po，every 3 weeks(q3w) ; Sintilimab at the dose 200mg，iv, d1, given every 3 weeks (q3w); Pemetrexed at the dose 500 mg/m2，iv，d1，given every 3 weeks (q3w); Carboplatin at the dose AUC=4~5，iv，d1；given every 3 weeks (q3w); Maintenance treatment：After 4~6 cycles of carboplatin treatment, Sintilimab 200mg, iv, d1, q3w；Fruquintinib RP2D intermittent(2 weeks on/1 weeks off), po，q3w； pemetrexed 500mg/m2, d1,iv, q3w until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal

SUMMARY:
A phase II study to assess the efficacy and safety of Fruquintinib Combined With Sintilimab and Chemotherapy as a first-line treatment in patients with unresectable or metastatic advanced Wild-type Genotype non-squamous Non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary provision of informed consent.
2. Males or females aged 18-75.
3. Histological or cytologically confirmed NSCLC, metastatic or non-resectable (stage IIIB-Ⅳ).
4. Not suitable for targeted therapy (patients with non-squamous NSCLC have no EGFR, ALK, gene mutation)
5. At least one lesion can be measured by imaging.
6. Have not received systemic treatment in the past.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
8. Life expectancy ≥ 12 weeks.
9. Female of childbearing age must have a negative pregnancy test (serum or urine) within 7 days before enrolment.

Exclusion Criteria:

1. Histological or cytologically confirmed small cell lung cancer (SCLC), including lung cancer mixed with SCLC and NSCLC.
2. Diagnosed with other malignant diseases other than NSCLC within 5 years.
3. Have participated in other interventional clinical research treatments now or within 4 weeks.
4. Have previously received multi-targeted kinase inhibitors therapy.
5. Have active autoimmune diseases requiring systemic treatment within 2 years.
6. Received systemic glucocorticoid therapy or immunosuppressive therapy within 2 weeks.
7. Clinically uncontrollable pleural effusion/abdominal effusion.
8. Vaccinated vaccines or attenuated vaccines within 4 weeks before the group;
9. Pregnant or breastfeeding females.
10. Other serious hazards to the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months
  To assess the efficacy of Fruquintinib Combined With Chemotherapy as second-

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 24 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate (DCR) | up to 24 months
  CR + PR + SD rate according to the RECIST
Overall Survival（OS） | up to 24 months
  Overall survival is determined from the date of treatment to death from any cause or the last follow-up date

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No